CLINICAL TRIAL: NCT03542825
Title: Outcome of Oral Lactoferrin in Comparison to Amino Acid Chelated Iron and Ferrous Sulphate Supplementation During Pregnancy: A Randomized Control Trial
Brief Title: Oral Lactoferrin Versus Iron Supplementation During Pregnancy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Mohammad Abdel-Rahman Mohammad Ahmed, Principal investigator, South Valley University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: OBGYN 003
Record Dates: First submitted 2018-05-20; First posted 2018-05-31 (Actual); Last update posted 2018-12-28 (Actual); Status verified 2018-12

CONDITIONS: Iron-deficiency
Keywords: Iron; Deficiency
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Lactoferrin; Iron-Dextran Complex; Iron Chelating Agents

STUDY DESIGN:
Intervention Model Description: 3 groups of pregnant women will be assigned for each intervention
Who Masked: Participant, Care Provider
Masking Description: Double blinded (participant and care giver)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Iron Sulphate (Active Comparator): ferrous sulphate 150 mg iron capsule once daily for 3 consecutive months.
  Interventions: Drug: Iron Supplement
- Amino acid Chelated (Active Comparator): amino acid chelated iron capsule 15mg for 3 consecutive months.
  Interventions: Drug: Chelates, Iron
- Lactoferrin (Active Comparator): lactoferrin 100 mg sachets once daily for 3 consecutive months.
  Interventions: Drug: Lactoferrin

INTERVENTIONS:
Drug: Lactoferrin — parallel use of the three drugs to compare the efficacy of each arm in prevention of anemia
  Arms: Lactoferrin
Drug: Iron Supplement — Iron Sulphate 150 mg once daily
  Other Names: Iron Sulphate
  Arms: Iron Sulphate
Drug: Chelates, Iron — Amino acid chelated iron capsules contain 15 mg
  Other Names: Amino acid chelated iron
  Arms: Amino acid Chelated

SUMMARY:
Iron deficiency anemia (IDA) is the condition in which there is anemia due to a lack of iron. The oral route is preferred to the parenteral route to replace iron stores [Sharma JB; et al., 2004]. Inorganic iron has poor bio-availability in addition to many side effects, including gastrointestinal discomfort, nausea, vomiting, diarrhea and constipation and it may sometimes increase susceptibility to infection [ So¨lvell L; et al., 1970].

DETAILED DESCRIPTION:
Iron deficiency anemia (IDA) is the condition in which there is anemia due to a lack of iron. The oral route is preferred to the parenteral route to replace iron stores. This allows the normal mechanism of absorption to be used, in addition to being an inexpensive and effective treatment [Sharma JB; et al., 2004]. Inorganic iron has poor bio-availability in addition to many side effects, including gastrointestinal discomfort, nausea, vomiting, diarrhea and constipation and it may sometimes increase susceptibility to infection [ So¨lvell L; et al., 1970].

Furthermore, routine iron supplementation has recently been challenged. The British Society for Hematology, Obstetric Hematology Group (BSH OHG) and the British Committee for Standards in Hematology (BCSH) recommend screening by Full blood count (FBC) at booking and at 28 weeks instead of universal iron supplementation [Pavord S. 2012]. Lactoferrin is a high-affinity cationic iron binding glycoprotein [Baker EN, 2005]. Bovine Lactoferrin is currently available pharmaceutical preparation. It is in to safe and effective in treating pregnant women suffering from ID and IDA [Mohamed Rezk, et al. 2015]. This study will compare the efficacy of these three available options.

ELIGIBILITY:
Inclusion Criteria:

• Pregnant women (aged 20-40 yrs.) with single fetus, in the second trimester, with normal haemoglobin level (Hb level ≥10.5 gm /dl) will be enrolled.

Exclusion Criteria:

* Women with anaemia (Hb level ≤10.5 gm. /dl) due to any causes, such as chronic blood loss, haemolytic anaemia and thalassemia (including thalassemia trait).
* History of peptic ulcer.
* Medical complications with pregnancy (such as cardiovascular, thyroid, pituitary, nutritional, renal, liver diseases, diabetes mellitus (DM) and hypertension (HTN).
* Fetal abnormalities such as microcephaly, intrauterine growth restriction (IUGR).

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 300 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-09-01 (Actual); Study Completion 2018-10-01 (Actual)

PRIMARY OUTCOMES:
change in haemoglobin level after 4 weeks of use. | 4 weeks
  difference in haemoglobin levelbetween before and after supplementation

SECONDARY OUTCOMES:
side effect profile | 4 weeks
  All women will be asked to keep a diary of five potential gastrointestinal side effects (Epigastric pain, nausea, vomiting, diarrhoea and constipation).

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad AM Ahmed, MD, Principal Investigator — South Valley University, Qena Faculty of Medicine, Obstetrics and Gynecology Department, Qena, Qena, Egypt
Locations (1):
- South Valley University, Qena Faculty of Medicine, Obstetrics and Gynecology Department, Qina, Qena Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared in unanonomous manner with the predetermined group of researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: throughout the period of research until end of the study
Access Criteria: IPD will be shared with the predetermined group of researchers as accepted by the local ethical and research committee.

REFERENCES:
- [Background] Sharma JB, Jain S, Mallika V, Singh T, Kumar A, Arora R, Murthy NS. A prospective, partially randomized study of pregnancy outcomes and hematologic responses to oral and intramuscular iron treatment in moderately anemic pregnant women. Am J Clin Nutr. 2004 Jan;79(1):116-22. doi: 10.1093/ajcn/79.1.116. PMID 14684407
- [Background] Pavord S, Myers B, Robinson S, Allard S, Strong J, Oppenheimer C; British Committee for Standards in Haematology. UK guidelines on the management of iron deficiency in pregnancy. Br J Haematol. 2012 Mar;156(5):588-600. doi: 10.1111/j.1365-2141.2011.09012.x. PMID 22512001
- [Background] Baker EN, Baker HM. Molecular structure, binding properties and dynamics of lactoferrin. Cell Mol Life Sci. 2005 Nov;62(22):2531-9. doi: 10.1007/s00018-005-5368-9. PMID 16261257
- [Background] Abu Hashim H, Foda O, Ghayaty E. Lactoferrin or ferrous salts for iron deficiency anemia in pregnancy: A meta-analysis of randomized trials. Eur J Obstet Gynecol Reprod Biol. 2017 Dec;219:45-52. doi: 10.1016/j.ejogrb.2017.10.003. Epub 2017 Oct 4. PMID 29059584